CLINICAL TRIAL: NCT03655587
Title: Impact of an Orthotic Intervention on Physical Function in Children With Chemotherapy-induced Peripheral Neuropathy
Brief Title: Impact of an Orthotic Intervention in Children With Peripheral Neuropathy
Acronym: IOPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Collaborators: Pine Tree Apple Tennis Classic Foundation (Unknown); St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1510-105
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Gait, Drop Foot; Chemotherapy-induced Peripheral Neuropathy; Acute Lymphocytic Leukemia, Pediatric; Rhabdomyosarcoma; Wilms Tumor
MeSH Terms: conditions — Gait Disorders, Neurologic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Rhabdomyosarcoma; Wilms Tumor

STUDY DESIGN:
Intervention Model Description: Each group gets one of the 2 types of orthotics.
Who Masked: Outcomes Assessor
Masking Description: Assessor blinded to the intervention type
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solid ankle foot orthotic (Experimental): This is a leg brace that is made to fit the contour of the patient's foot, ankle, and lower leg. The two pull solid ankle AFO is fabricated from a rigid polypropylene outer boot and a more flexible silicone inner boot. It is commonly used in rehabilitation to improve gait in pediatric and adult populations. A certified orthotist fabricates the device. This device is lawfully marketed in the United States. It is not regulated by the FDA.
  Interventions: Device: Solid ankle foot orthotic
- Resting night splint (Active Comparator): An ankle resting night spring (RNS) is an off-the-shelf device that provides static sagittal plane dorsiflexion. The RNS is worn nocturnally to provide maximal stretch/length to the gastrocsoleus to maintain or increase dorsiflexion ROM and/or to prevent further regressions in ankle range. It is not regulated by the FDA.
  Interventions: Device: Resting night splint

INTERVENTIONS:
Device: Solid ankle foot orthotic
  Arms: Solid ankle foot orthotic
Device: Resting night splint
  Arms: Resting night splint

SUMMARY:
This research study will investigate the effect of two orthotic (brace) devices for the ankle and foot on walking and ankle flexibility in children with cancer not involving the brain or spinal cord.

DETAILED DESCRIPTION:
This research study will investigate the effect of two orthotic (brace) devices for the ankle and foot on walking and ankle flexibility in children with cancer not involving the brain or spinal cord. Children undergoing treatment for cancer can suffer from decreased flexibility, strength, balance and endurance from the cancer and from direct effects of the chemotherapy agents. These impairments have been shown to continue years after treatment end, with adult survivors of cancer being less physically active than their siblings. Children, whose chemotherapy includes vincristine, can develop damage to their peripheral nervous system affecting the strength, sensation, and flexibility in their hands and feet. This can then lead to a change in their walking pattern and ankle flexibility and likely contributes to decreased physical activity level and fatigue.

In our clinical practice and pilot work, we know that solid ankle orthotics can be effective in improving gait quality and ankle flexibility. However, in other areas of the country, researchers have published on the effectiveness of using a different type of brace, called a resting night splint, to improve gait and ankle function. Thus, we are studying the comparative efficacy of these two approaches.

Our published pilot study demonstrated that children with cancer were able to wear solid ankle orthotics without an impact on their safety. This study will further the research by comparing the effect of the solid ankle foot orthotic against a resting splint worn at night on walking and ankle flexibility in children with cancer.

Ankle foot orthotics improve a walking pattern by positioning the foot and ankle so that the toe can clear the floor more easily and the child can take a longer step. This decreases the energy needed for a child to walk, allowing the ability to walk longer distances or increase physical activity level. The AFO will also increase ankle flexibility by stretching the muscle while walking. If the child or adolescent walks with an increased step length, they will give a greater stretch to the calf muscles while walking. In contrast, the resting night splint can increase ankle flexibility by providing a gentle stretch to the calf muscles while sleeping, therefore allowing improved ankle movement when walking and a longer step length. We will examine the impact of these orthotics on walking, ankle flexibility, ankle strength, aerobic capacity, self-reported fatigue, as well as the ability of the children to wear the orthotic as prescribed and the severity of the damage to the nervous system.

Children and adolescents who are found to have ankle weakness, ankle tightness, and damage to their peripheral nervous system as a result of cancer treatment will be referred to the study by the treating physical therapist (PT). The PT will contact the investigators and they will invite the child or adolescent to participate in the study. Using previously established measurements in children with cancer, we will measure walking pattern, ankle strength, ankle flexibility, foot posture, level of physical activity, and level of fatigue prior to the orthotic intervention. The subject will then be randomized between an 8-week AFO or RNS intervention. The orthotic will be made with a small temperature sensor that will collect data on wearing time of the brace. After 8 weeks of orthotic wear, we will repeat the measurements and compare results between the two orthotic types.

ELIGIBILITY:
Inclusion Criteria:

* 1)between 5-14 years of age; 2)demonstrated neuropathy as evidenced by a Ped-mTNS score>4; 3)normalized step length more than 1 standard deviation below mean for age26 ; 4)ankle DF PROM <10 degrees ; 5) able to give assent according to institutional guidelines; and 6) have parental consent to participate.

Exclusion Criteria:

* 1)lower extremity sarcomas; 2) central nervous system tumors; 3) an antecedent neurological, developmental, or genetic disorder; and 4)osteonecrosis (ON) 5)Less than antigravity dorsiflexion strength 6) neuroblastoma

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Step length | 8 weeks
  Length of the step in participant's gait measured by the gaitrite analysis system

SECONDARY OUTCOMES:
Ankle range of motion | 8 weeks
  Passive and active ankle dorsiflexion measured by goniometry
Ankle strength | 8 weeks
  Ankle dorsiflexion and plantarflexion strength measured by dynamometer
Gait capacity | 8 weeks
  Measured by the 6-minute walk test distance
Foot posture | 8 weeks
  Measured by the foot posture index

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Tanner, MPT, Principal Investigator — Children's Minnesota
Locations (2):
- United States (2):
  - Children's Minnesota, Minneapolis, Minnesota
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No